CLINICAL TRIAL: NCT01978158
Title: Effects of Oxygen Status on Endotoxemia Induced Inflammation and Hypoxia Inducible Factor-1α. A Pilot Proof of Principle Study
Brief Title: Effects of Oxygen Status on Endotoxemia Induced Inflammation and Hypoxia Inducible Factor-1α
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OX2; 2013-002390-21 (EudraCT Number); NL44630.091.13 (Other: CCMO); 2013/290 (Other: CMO Arnhem-Nijmegen)
Record Dates: First submitted 2013-10-31; First posted 2013-11-07 (Estimated); Last update posted 2015-05-20 (Estimated); Status verified 2015-05

CONDITIONS: Hypoxia; Normoxia; Hyperoxia
Keywords: Oxygen; Hypoxia; Hyperoxia; Inflammation; Innate immunity
MeSH Terms: conditions — Hypoxia; Hyperoxia; Inflammation | interventions — Lipopolysaccharides

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Hypoxia (Experimental): Subjects will be breathing an individualized mix of nitrogen and room air titrated to an oxygen saturation of 80-85%.
  Interventions: Drug: Lipopolysaccharide
- Hyperoxia (Experimental): Subjects will be breathing 100% of oxygen
  Interventions: Drug: Lipopolysaccharide
- Normoxia (Active Comparator): Subjects wil be breathing room air (21%)
  Interventions: Drug: Lipopolysaccharide

INTERVENTIONS:
Drug: Lipopolysaccharide — LPS is used to elicit an inflammatory response in all subjects
  Other Names: Purified LPS from Escherischa coli (O:113)

SUMMARY:
Oxygen is a widely available gas that is cheap, easy to get and extensively used in medicine. From animal studies it has become apparent that increasing or lowering the degree of oxygen in the blood, the inflammatory response can be altered. We will investigate of this is also true in humans by increasing, lowering or keeping oxygen levels normal while giving healthy subjects a short inflammatory stimulus.

DETAILED DESCRIPTION:
The primary objective of the study is to determine the effects of hyperoxia and hypoxia compared to normoxia in the human endotoxemia model on the innate immune reponse in healthy volunteers.

A parallel, randomized study in healthy male volunteers. The subjects will be randomized to hypoxia, hyperoxia, or normoxia, and will all undergo experimental human endotoxemia (administration of 2 ng/kg LPS iv).

In the hypoxia group: the subjects will breathe an individualized mix of nitrogen and room air for 3.5 hours using an air-tight respiratory helmet. The gas mixture will be adjusted to achieve a saturation of 80-85%. In the hyperoxia group, subjects will breathe 100% oxygen for 3.5 hours using the same respiratory helmet. In the normoxia group, subjects will breathe room air (21% oxygen, 79% nitrogen) also wearing the respiratory helmet. 1 hour after oxygen status adjustment (t=0), all subject will be administered an intravenous bolus (2ng/kg) of LPS derived from E coli O:113. 2.5 hours after LPS administration, the helmets will be removed and all subjects will breathe ambient room air.

The primary study endpoint is the difference in plasma cytokines between the hypoxia and normoxia group, and between the hyperoxia and normoxia group. Secondary objectives include HIF-1α protein and mRNA, aHIF mRNA expression in circulating leukocytes, measures of ROS, leukocyte phagocytosis, and cytokine production by leukocytes stimulated ex vivo with various inflammatory stimuli, and measurement of basic hemodynamic and ventilatory parameters and temperature.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent to participate in this trial
* Male subjects aged 18 to 35 years inclusive
* Healthy as determined by medical history, physical examination, vital signs, 12-lead electrocardiogram, and clinical laboratory parameters

Exclusion Criteria:

* Use of any medication(including herbal remedies and vitamin/mineral supplements) or recreational drugs within 7 days prior to profiling day
* Smoking
* Use of caffeine, or alcohol or within 1 day prior to profiling day
* Previous participation in a trial where LPS was administered
* Surgery or trauma with significant blood loss or blood donation within 3 months prior to profiling day
* Participation in another clinical trial within 3 months prior to profiling day.
* History, signs or symptoms of cardiovascular disease
* An implant that in the opinion of the investigator may make invasive procedures risky for the subject due to the increased risks associated with a possible infection.
* Subject has an implanted active cardiac device (ICD, IPG and/or CRT) Implanted active neurostimulation device
* Subject has internal jugular vein that cannot be accessed
* History of vaso-vagal collapse or of orthostatic hypotension
* History of atrial or ventricular arrhythmia
* Resting pulse rate ≤45 or ≥100 beats / min
* Hypertension (RR systolic >160 or RR diastolic >90)
* Hypotension (RR systolic <100 or RR diastolic <50)
* Conduction abnormalities on the ECG consisting of a 1st degree atrioventricular block or a complex bundle branch block
* Subject is diagnosed with epilepsy or history of seizures
* Renal impairment: plasma creatinine >120 μmol/L
* Liver function abnormality: alkaline phosphatase>230 U/L and/or ALT>90 U/L
* Coagulation abnormalities: APTT or PT > 1.5 times the reference range
* History of asthma
* Immuno-deficiency CRP > 20 mg/L, WBC > 12x109/L, or clinically significant acute illness, including infections, within 2 weeks before profiling day
* Known or suspected of not being able to comply with the trial protocol - Inability to personally provide written informed consent (e.g. for linguistic or mental reasons) and/or take part in the study.

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2013-10; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Plasma TNF-alpha concentration following LPS administration | 1 day
  Plasma TNF-α concentration after LPS administration (Area Under Curve); comparison of subjects treated with hypoxia compared to normoxia and hyperoxia compared to hypoxia

SECONDARY OUTCOMES:
Hypoxia Inducible Factor 1 alpha in circulating leukocytes | 1 day
  Hypoxia Inducible Factor 1 alpha in circulating neutrophils, lymfocytes and monocytes as measured with flow cytometry
Hypoxia Inducible Factor mRNA and anti Hypoxia Inducible Factor mRNA in circulating leukocytes | 24 hours
Reactive Oxygen Species in circulating leukocytes | 1 day
Phagocytic function of circulating leukocytes | 1 day
cytokine production after ex vivo stimulation of leukocytes | 1 day
circulating cytokines (including but not limited to IL-6, IL-10, IL-1RA) | 1 day
Hemodynamic parameters | 1 day
  Blood pressure, heart frequency, cardiac output measurement
ventilatory response | 1 day
  Measures of ventilation: respiratory rate, blood gas changes
adenosine metabolism | 1 day
  urine and plasma adenosine,adenosine receptor mRNA, purines
alkaline phosphatase | 1 day
cognitive function | 1 day
  neuropsychologic assessment of cognitive function
Hepcidin and iron parameters | 1 day
catecholamines and cortisol | 1 day
  adrenaline, noradrenaline, dopamine and cortisol
Neutrophilic function | 1 day
body temperature | 1 day
oxygen saturation and arterial blood gas | 1
subjective symptom scores | 1 day
high sensitive troponine | 1 day
iFABP | 1 day
brain specific proteins | 1 day
endocan | 1 day
downstream targets of HIF | 1 day
  adrenomedullin, VEGF, EPO
heart rate variability | 1 day
kidney injury markers in plasma and urine | 2 days
microbiome in feces | -1 day untill 1 week
markers of immunoparalysis | 1 day
  monocytic histone 3 lysine 4 trimethylation of the promotor region of pro-inflammatory genes, ex viv production of proinflammatory cytokines, HLA-DR expression on moncytes.
measures of coagulation and plateletfunction | 1 day
  platelet activation and platelet function, thrombin generation and other coagulation parameters, hematolocial infection profile using hematology analyser
meausures of coagulation and fibrinolysis | 1 day
  thrombin generation, thrombocyte function, ROTEM, plasmatic coagulation, fibrinolysis parameters

CONTACTS AND LOCATIONS:
Overall Officials: Peter Pickkers, MD, PhD, Principal Investigator — Intensive Care Medicine, Radboud University Nijmegen Medical Centre
Locations (1):
- Intensive Care Medicine, Nijmegen, Gelderland, Netherlands